CLINICAL TRIAL: NCT03719625
Title: Norepinephrine Versus Ephedrin for Prevention of Post Spinal Anesthesia in Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Head of the anesthesia intensive care department, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: prophylactic vasopressors
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-10

CONDITIONS: Maternal Hypotension Syndrome; Cesarean
MeSH Terms: interventions — Ephedrine; Norepinephrine

STUDY DESIGN:
Intervention Model Description: controlled, prospective, randomised trial comparing 2 interventions
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- norepinephrin group (Experimental): The patients of this group will recieve 0.5 micro gr/kg of norepinephin intravenously, the infusion will start during the intrathecal injection and during 10 minutes
  Interventions: Drug: Norepinephrine
- Ephedrin group (Experimental): The patients of this group will recieve 0,3mg/kg of Ephedrin intravenously, the infusion will start during the intrathecal injection and during 10 minutes
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Ephedrine — Comparaison of Norepinephrin and Ephedrin for prevention of the post spinal anesthesia in cesarean section
  Other Names: Ephedrin
  Arms: Ephedrin group
Drug: Norepinephrine — Comparaison of Norepinephrin and Ephedrin for prevention of the post spinal anesthesia in cesarean section
  Arms: norepinephrin group

SUMMARY:
Spinal anesthesia is still the gold standard anesthetic method for elective and urgent cesarean section, the post spinal hypotension remains the most frequent complication of this procedure and is still responsible of considerable maternel and fetal morbidity. It is recommanded to prevent this post spinal hypotension with fluid coloading and prophylactic vasopressors administration.

The aim of this study is to compare the efficency and the safety of norepinephrin and ephedrin prophylactic administration to reduce the incidence of post spinal hypotension in cesarean section.

DETAILED DESCRIPTION:
Spinal anesthesia is still the gold standard anesthetic method for elective and urgent cesarean section, the post spinal hypotension remains the most frequent complication of this procedure and is still responsible of considerable maternel and fetal morbidity. It is recommanded to prevent this post spinal hypotension with fluid coloading and prophylactic vasopressors administration. The prophylactic use of norepinephrin and phenylephrin has been validated by several studies, but few data are published concerning the comparaison between norepinephrin and ephedrine as preventive vasopressors in cesarean section; these molecules act on alpha and beta adrenergic receptors and could provide better maternal hemodynamics in parturients undergoing cesarean section under spinal anesthesia.

The aim of this study is to compare the efficency and the safety of norepinephrin and ephedrin prophylactic administration to reduce the incidence of post spinal hypotension in cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* full termed parturients scheduled for elective or semi urgent cesarean section under spinal anesthesia
* AGE>15 years
* ASA II status
* No history of hypertension, preeclampsia or cardiopathy
* BMI<40

Exclusion Criteria:

* cesarean section under genearl anesthesia or epidural analgesia during labor

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — this study is exclusively including paturients undergoing cesarean section
Enrollment: 200 (Estimated)
Dates: Start 2019-01-02 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of post spinal hypotension | during the first 20 minutes after spinal anesthesia
  decrease of systolic arterial blood pressure > 20% baseline

SECONDARY OUTCOMES:
Lowest systolic blood pressure | uring the first 20 minutes after spinal anesthesia
  Lowest systolic blood pressure recorded after spinal anesthesia
Incidence of bradycardia | during the first 20 minutes after spinal anesthesia
  heart rate<50 beats/min
incidence of nausea and/or vomiting | during the first 20 minutes after spinal anesthesia
  incidence of nausea and/or vomiting
Apgar score | 20min after spinal anesthesia
  Apgar score at 1 min, 5 min, 10 min
fetal ph | 20min after spinal anesthesia
  fetal ph
fetal blood lactates | 20min after spinal anesthesia
  fetal blood lactates

IPD SHARING:
Plan to Share IPD: Undecided